CLINICAL TRIAL: NCT00492726
Title: A Prospective, Randomized, Double-dummy, Double-blind, Multicenter Trial Comparing the Safety and Efficacy of Intravenous Moxifloxacin 400 mg IV QD 24 Hours to That of Ertapenem 1.0 g IV QD 24 Hours for 5 to 14 Days for the Treatment of Subjects With Complicated Intra-abdominal Infections (PROMISE Study)
Brief Title: Therapy of Complicated Intra-Abdominal Infections With Moxifloxacin or Ertapenem
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11976; 2006-000874-56 (EudraCT Number)
Record Dates: First submitted 2007-06-26; First posted 2007-06-27 (Estimated); Results first posted 2010-03-03 (Estimated); Last update posted 2014-11-07 (Estimated); Status verified 2014-11

CONDITIONS: Infection
Keywords: Complicated Intra-Abdominal Infections
MeSH Terms: conditions — Infections | interventions — Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Moxifloxacin (Avelox, BAY12-8039) (Experimental): Subjects received placebo matching the comparator (Ertapenem dummy) and Moxifloxacin 400 mg in 250 mL for intravenous infusion every 24 hours.
  Interventions: Drug: Moxifloxacin (Avelox, BAY12-8039)
- Ertapenem (Active Comparator): Subject received Ertapenem 1.0 g in 50 mL for intravenous infusion and placebo matching Moxifloxacin (Moxifloxacin dummy) every 24 hours.
  Interventions: Drug: Ertapenem intravenous

INTERVENTIONS:
Drug: Moxifloxacin (Avelox, BAY12-8039) — Moxifloxacin, 400mg, administered intravenously once daily
  Arms: Moxifloxacin (Avelox, BAY12-8039)
Drug: Ertapenem intravenous — Active treatment: Ertapenem 1.0g, administered intravenously once daily
  Arms: Ertapenem

SUMMARY:
A study to compare the safety and efficacy of moxifloxacin to ertapenem in patients with intra-abdominal infections.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized men or women >/=18 years of age
* Expected duration of treatment with intravenous antibiotics anticipated to be >/= 5 full days but not exceeding 14 days
* Ability to provide documented and signed written informed consent
* Confirmed or suspected intra abdominal infection defined as follows:

  * For a confirmed intra abdominal infection, a surgical procedure (laparotomy or laparoscopy) must have been performed within 24 hours prior to enrollment and reveal at least one of the following:

    * Gross peritoneal inflammation with purulent exudates (i.e. peritonitis)
    * Intra abdominal abscess
    * Macroscopic intestinal perforation with localized or diffuse peritonitis
* Subjects enrolled on the basis of a suspected intra abdominal infection must have:

  * Radiological evidence [abdominal plain films, computed tomography (CT), magnetic resonance imaging (MRI) or ultrasound] of gastrointestinal perforation or intra-abdominal abscess and the following signs and symptoms:

    * Symptoms referable to the abdominal cavity (e.g. anorexia, nausea, vomiting or pain), lasting for at least 24 hours
    * Tenderness (with or without rebound), involuntary guarding, absent or diminished bowel sounds, or abdominal wall rigidity
  * At least two of the following SIRS criteria:

    * Temperature > 38.0°C rectal or tympanic membrane, or temperature < 36.0°C rectal or tympanic
    * Heart rate > 90/min
    * Respiratory rate > 20/min
    * WBC >12,000 cells/mm3 or < 4,000 cells/ mm3
  * The subject must be scheduled for a surgical procedure (laparotomy or laparoscopy) within 24 hours of enrollment of the study

Exclusion Criteria:

* Known hypersensitivity to quinolones, and/or to carbapenems and/or to any other type of beta lactam antibiotic drugs (e.g. penicillins or cephalosporins), or any of the excipients
* Women who are pregnant or lactating or in whom pregnancy cannot be excluded
* History of tendon disease/disorder related to quinolone treatment
* Known congenital or documented acquired QT prolongation; uncorrected hypokalemia; clinically relevant bradycardia; clinically relevant heart failure with reduced left ventricular ejection fraction; previous history of symptomatic arrhythmias
* Concomitant use of any of the following drugs, reported to increase the QT interval: antiarrhythmics class IA (e.g. quinidine, hydroquinidine, disopyramide) or antiarrhythmics class III (e.g., amiodarone, sotalol, dofetilide, ibutilide), neuroleptics (e.g. phenothiazines, pimozide, sertindole, haloperidol, sultopride), tricyclic antidepressive agents, certain antimicrobials (sparfloxacin, erythromycin IV, pentamidine, antimalarials, particularly halofantrine), certain antihistaminics (terfenadine, astemizole, mizolastine), and others (cisapride, vincamine IV, bepridil, diphemanil)
* Known severe end stage liver disease
* Creatinine clearance </= 30 mL/min/1.73 m2
* Systemic antibacterial therapy administered for more than 24 hours within 7 days of enrollment
* Need for systemic antibacterial therapy with agents other than those described in the study protocol
* Indwelling peritoneal catheter
* Pre existing ascites and presumed spontaneous bacterial peritonitis
* Perforation of the stomach or duodenum, if the duration of perforation is less than 24 hours or if operated on within 24 hours of perforation
* Perforation of the small bowel (excluding the duodenum) or large bowel, if the duration of perforation is less than 12 hours or if operated on within 12 hours of perforation
* All pancreatic processes including pancreatic sepsis, peri-pancreatic sepsis, or an intra abdominal infection secondary to pancreatitis
* Liver and splenic abscess
* Transmural bowel ischemia or necrosis without perforation or established peritonitis or abscess
* Acute and gangrenous cholecystitis without perforation
* Acute cholangitis
* Early acute, suppurative, or gangrenous non-perforated appendicitis
* Subjects requiring antibiotic irrigations of the abdominal cavity or surgical wound
* Treatment with "open abdomen" or marsupialization, or multiple planned re laparotomies
* Infections originating from the female genital tract
* Peri-nephric infections
* Evidence of sepsis with shock requiring the administration of vasopressors for more than 4 consecutive hours
* Known rapidly fatal underlying disease (death expected within 6 months)
* Neutropenia (neutrophil count < 1,000/mL) caused by immunosuppressive therapy or malignancy
* Receiving chronic treatment with known immunosuppressant therapy (including chronic treatment with > 15 mg/day of systemic prednisone or equivalent)
* Subjects known to have AIDS (CD4 count < 200/mL) or HIV seropositives who are receiving HAART (HIV positive subjects may be included. HIV testing is not required for this study protocol)
* Subjects with a malignant or pre malignant hematological condition, including Hodgkin's disease and non-Hodgkin lymphoma (subjects with solid tumor can be included in the study)
* Subjects with a Body Mass Index >/= 45 kg/m2
* Previous enrollment in this study
* Participation in any clinical investigational drug study within the previous 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 804 (Actual)
Dates: Start 2006-07; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (47):
- Argentina (9):
  - Ciudadela, Buenos Aires
  - De Febrero 3, Buenos Aires
  - Merlo, Buenos Aires
  - San Juan Bautista, Buenos Aires
  - Buenos Aires, Ciudad Auton. de Buenos Aires
  - Córdoba, Córdoba Province
  - Mendoza, Mendoza Province
  - Rosario, Santa Fe Province
  - Capital Federal
- Belgium (2):
  - Bruxelles - Brussel
  - Ghent
- Bulgaria (3):
  - Pleven
  - Rousse
  - Sofia
- Estonia (3):
  - Kohtla-Järve
  - Tallinn
  - Tartu
- France (2):
  - Amilly
  - Besançon
- Germany (5):
  - Heidelberg, Baden-Wurttemberg
  - Beeskow, Brandenburg
  - Hanover, Lower Saxony
  - Paderborn, North Rhine-Westphalia
  - Homburg, Saarland
- Rio Patras, Greece
- Israel (2):
  - Haifa
  - Kfar Saba
- Latvia (5):
  - Daugavpils
  - Liepāja
  - Rēzekne
  - Riga
  - Valmiera
- Lithuania (3):
  - Kaunas
  - Klaipėda
  - Vilnius
- Romania (5):
  - Brasov
  - Bucharest
  - Cluj-Napoca
  - Oradea
  - Timișoara
- Russia (2):
  - Moscow
  - Smolensk
- South Africa (3):
  - Cape Town, Cape
  - Pretoria, Gauteng
  - Somerset West, Western Cape
- Spain (2):
  - L'Hospitalet de Llobregat, Barcelona
  - Madrid, Madrid

REFERENCES:
- [Result] De Waele JJ, Tellado JM, Alder J, Reimnitz P, Jensen M, Hampel B, Arvis P. Randomised clinical trial of moxifloxacin versus ertapenem in complicated intra-abdominal infections: results of the PROMISE study. Int J Antimicrob Agents. 2013 Jan;41(1):57-64. doi: 10.1016/j.ijantimicag.2012.08.013. Epub 2012 Nov 13. PMID 23153963
- See also: Click here and search for information of Bayer products for Europe — http://www.clinicaltrialsregister.eu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled from 02 July 2006 to 31 December 2008 at 52 centers in 14 countries: Argentina (9), Belgium (3), Bulgaria (4), Estonia (3), France (2 ), Germany (5), Greece (1), Israel (2), Latvia (6), Lithuania (4), Romania (5), Russia (3), South Africa (3), and Spain (2).
Pre-assignment Details: 830 subjects screened, 804 randomized. 6 not treated. Safety/Intent to treat population = 798 subjects with at least 1 dose taken and 1 observation after intake (Moxifloxacin 408; Ertapenem 390). Per protocol population = 699 subjects with no major protocol deviations that would have influenced the primary outcome (Moxifloxacin 352; Ertapenem 347).
Period: Overall Study
Arm/Group | Moxifloxacin (Avelox, BAY12-8039) | Ertapenem
Started | 410 | 394
End of Treatment (EOT, Day 5 to 14) | 387 | 377
End of Study | 360 | 358
Completed | 360 | 358
Not Completed | 50 | 36
Not completed — Adverse Event | 10 | 6
Not completed — Death | 7 | 2
Not completed — Lack of Efficacy | 0 | 2
Not completed — Lost to Follow-up | 27 | 19
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 6 | 3
Not completed — Non compliant with study medication | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Moxifloxacin (Avelox, BAY12-8039) | Ertapenem | Total
Number analyzed (Participants) | 410 | 394 | 804
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.1 (18.3) | 47.0 (18.2) | 47.4 (18.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 156 | 131 | 287
  Male | 254 | 263 | 517

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Achieving Clinical Cure at Test of Cure (TOC) Visit in the Per Protocol Population
Description: Clinical cure at TOC = resolution or improvement of clinical signs and symptoms related to the infection without the occurrence of a wound infection requiring a systemic antibiotic treatment. Clinical failure at TOC = either failure to respond or insufficient lessening of the signs and symptoms of infection at end of treatment (EOT) or reappearance of the signs and symptoms of the original infection from EOT up to TOC or wound infection requiring additional systemic antimicrobial therapy at any time up to TOC.
Time Frame: 21 to 28 days after completion of study drug therapy
Population: The per protocol population was the main analysis set for the assessment of clinical response and was defined as those subjects with no major protocol deviations that would have influenced the primary outcome.
Measure: Number; unit: participants
Arm/Group | Moxifloxacin (Avelox, BAY12-8039) | Ertapenem
Number analyzed (Participants) | 352 | 347
participants
  Clinical Cure | 315 | 324
  Clinical Failure | 37 | 23
Statistical Analysis 1: Comparison: Moxifloxacin (Avelox, BAY12-8039) vs Ertapenem; Calculated were 95% confidence intervals for the difference in success rates between treatment groups (moxifloxacin minus comparator); Test type: Non-Inferiority or Equivalence — The non-inferiority margin was set to 10% in the protocol, in agreement with FDA recommendations. Sample size was estimated using the method as described in Farrington-Manning. Estimation was performed to achieve 85% power, based on the equivalence delta of 10%, and a clinical success rate of 80% in the per protocol population; Difference of cure rates (in percent) = -3.8, 95% CI [-7.9 to 0.4] — A positive value indicates an advantage for the treatment group of moxifloxacin, a negative value an advantage for the comparator group

2. Secondary Outcome: Number of Subjects Achieving Clinical Improvement During Treatment in the Per Protocol Population
Description: Clinical improvement = Reduction in the severity and/or number of signs and symptoms of infection.Clinical failure = Failure to respond/insufficient lessening of signs and symptoms of infection requiring a modification/addition of antibacterial therapy, or a second surgical intervention (unless the original surgery was deemed inadequate). Development of a wound infection requiring alternative/additional antibiotic therapy was considered a failure. Failed subjects must have had 3 full days of therapy administered.
Time Frame: During treatment at day 5 +/- 1 day
Population: Per protocol population comprising subjects with no major protocol deviations that would have influenced the primary outcome.
Measure: Number; unit: participants
Arm/Group | Moxifloxacin (Avelox, BAY12-8039) | Ertapenem
Number analyzed (Participants) | 352 | 347
participants
  Clinical Improvement | 210 | 194
  Clinical Failure | 0 | 2
  Missing | 142 | 151
Statistical Analysis 1: Comparison: Moxifloxacin (Avelox, BAY12-8039) vs Ertapenem; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Sample size estimation was based on the primary efficacy variable; Difference in improvement rates (in %) = 1.1, 95% CI [-0.4 to 2.7] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Number of Subjects Achieving Bacteriological Success During Treatment in the Per Protocol Population With Causative Organism(s)
Description: Bacteriological success = response classified as 'eradication' or 'presumed eradication' without occurrence of a superinfection. Bacteriological failure = response classified as 'persistence', 'presumed persistence', or 'superinfection'.
Time Frame: During treatment at day 5 +/- 1 day
Population: Per protocol population (subjects with no major protocol deviations that would have influenced the primary outcome) with causative organism(s).
Measure: Number; unit: participants
Arm/Group | Moxifloxacin (Avelox, BAY12-8039) | Ertapenem
Number analyzed (Participants) | 297 | 276
participants
  Eradication | 5 | 5
  Presumed Eradication | 170 | 149
  Persistence | 16 | 7
  Presumed Persistence | 0 | 2
  Superinfections | 0 | 1
Statistical Analysis 1: Comparison: Moxifloxacin (Avelox, BAY12-8039) vs Ertapenem; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Sample size estimation was based on the primary efficacy variable; Difference in bact. success rates (in %) = -3.9, 95% CI [-8.8 to 1.0] — A positive value indicates an advantage for the treatment group of moxifloxacin, a negative value an advantage for the comparator group. Presumed eradications and eradications without superinfection were considered bacteriological successes

4. Secondary Outcome: Number of Subjects Achieving Clinical Cure at End of Therapy (EOT) Visit in the Per Protocol Population
Description: Clinical cure = resolution/improvement of clinical signs and symptoms related to the infection without wound infection requiring systemic antibiotic treatment. Clinical failure = Failure to respond/insufficient lessening of signs and symptoms of infection requiring a modification/addition of antibacterial therapy, or a second surgical intervention (unless the original surgery was deemed inadequate). Development of a wound infection requiring alternative/additional antibiotic therapy was considered a failure. Failed subjects must have had 3 full days of therapy administered.
Time Frame: after 5 - 14 days of therapy
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Moxifloxacin (Avelox, BAY12-8039) | Ertapenem
Number analyzed (Participants) | 352 | 347
participants
  Clinical Cure | 328 | 330
  Clinical Failure | 23 | 17
  Missing | 1 | 0
Statistical Analysis 1: Comparison: Moxifloxacin (Avelox, BAY12-8039) vs Ertapenem; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Sample size estimation was based on the primary efficacy variable; Difference of cure rates (in percent) = -1.5, 95% CI [-5.0 to 1.9] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Number of Subjects Achieving Bacteriological Success at EOT Visit in the Per Protocol Population With Causative Organism(s)
Description: as for outcome 3
Time Frame: After 5 - 14 days of therapy
Population: Per protocol population (subjects with no major protocol deviations that would have influenced the primary outcome) with causative organism(s). For one patient in the Moxifloxacin group, the data is missing due to missing EOT visit (not displayed in the table below).
Measure: Number; unit: participants
Arm/Group | Moxifloxacin (Avelox, BAY12-8039) | Ertapenem
Number analyzed (Participants) | 297 | 276
participants
  Eradication | 5 | 7
  Presumed Eradication | 257 | 247
  Persistence | 20 | 9
  Presumed Persistence | 13 | 11
  Superinfections | 1 | 2
  Indeterminate/missing | 1 | 0
Statistical Analysis 1: Comparison: Moxifloxacin (Avelox, BAY12-8039) vs Ertapenem; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Sample size estimation was based on the primary efficacy variable; Difference in bact. success rates (in %) = -3.9, 95% CI [-8.8 to 1.0] — [estimate comment as in outcome 3, analysis 1]

6. Secondary Outcome: Number of Subjects Achieving Bacteriological Success at TOC Visit in the Per Protocol Population With Causative Organism(s)
Description: Bacteriological success = response classified as 'eradication' or 'presumed eradication' without occurrence of a superinfection. Bacteriological failure = response classified as 'persistence', 'presumed persistence', or 'superinfection' - additionally, any recurrence or reinfection was treated as bacteriological failure at TOC.
Time Frame: 21 - 28 days after end of therapy
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Moxifloxacin (Avelox, BAY12-8039) | Ertapenem
Number analyzed (Participants) | 297 | 276
participants
  Eradication | 0 | 0
  Presumed Eradication | 257 | 249
  Persistence | 20 | 9
  Presumed Persistence | 20 | 18
  Superinfections | 0 | 0
  Reinfections | 0 | 0
Statistical Analysis 1: Comparison: Moxifloxacin (Avelox, BAY12-8039) vs Ertapenem; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Sample size estimation was based on the primary efficacy variable; Difference in bact. success rates (in %) = -3.8, 95% CI [-9.0 to 1.5] — A positive value indicates an advantage for the treatment group of moxifloxacin, a negative value an advantage for the comparator group. Presumed eradications and eradications without super- or reinfection were considered bacteriological successes

7. Secondary Outcome: Number of Subjects Achieving Clinical Cure at TOC Visit in the Per Protocol Population With Causative Organism(s)
Description: as for outcome 1
Time Frame: 21 - 28 days after end of therapy
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Moxifloxacin (Avelox, BAY12-8039) | Ertapenem
Number analyzed (Participants) | 297 | 276
participants
  Clinical Cure | 265 | 254
  Clinical Failure | 32 | 22
Statistical Analysis 1: Comparison: Moxifloxacin (Avelox, BAY12-8039) vs Ertapenem; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Sample size estimation was based on the primary efficacy variable; Difference of cure rates (in percent) = -2.9, 95% CI [-7.6 to 1.9] — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Number of Subjects Who Died Due to Intra-abdominal Infections
Description: Number of subjects who had died due to intra abdominal infections by the time of TOC visit.
Time Frame: 21 - 28 days after end of treatment at TOC Visit
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Moxifloxacin (Avelox, BAY12-8039) | Ertapenem
Number analyzed (Participants) | 352 | 347
participants
  Yes | 3 | 1
  No | 349 | 346

9. Secondary Outcome: Duration of Hospitalization
Description: Duration of hospitalization in the per protocol population.
Time Frame: From the first admission date to the discharge date (from 4 to 71 days after start of study medication)
Population: Numbers refer to patients in the per protocol population with known end of hospitalization date.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Moxifloxacin (Avelox, BAY12-8039) | Ertapenem
Number analyzed (Participants) | 346 | 343
days | 11.7 (7.3) | 11.2 (7.8)

10. Secondary Outcome: Duration of Hospitalization Postoperatively
Description: Duration of hospitalization after the first surgery until discharge in the per protocol population.
Time Frame: Duration of hospitalization after the first surgery until discharge date (from 4 to 71 days after start of study medication)
Population: Numbers refer to patients in the per protocol population with known end of hospitalization date.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Moxifloxacin (Avelox, BAY12-8039) | Ertapenem
Number analyzed (Participants) | 346 | 343
days | 11.1 (7.1) | 10.7 (7.2)

ADVERSE EVENTS:
Arm/Group | Moxifloxacin (Avelox, BAY12-8039) | Ertapenem
Serious Adverse Events (participants affected / at risk) | 60/408 | 48/390
Other Adverse Events (participants affected / at risk) | 115/408 | 87/390
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Moxifloxacin (Avelox, BAY12-8039) (N=408) | Ertapenem (N=390)
Acute mycardial infarction (Cardiac disorders) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 7 (7) | 2 (3)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 2 (2) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tachyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 0 (0)
Colonic fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal fistula (Gastrointestinal disorders) | 1 (1) | 3 (4)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peritonitis (Gastrointestinal disorders) | 3 (3) | 2 (2)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mechanical ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Jejunal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Impaired healing (General disorders) | 1 (1) | 0 (0)
Multi-organ failure (General disorders) | 4 (4) | 2 (2)
Unevaluable event (General disorders) | 4 (4) | 2 (2)
Acute hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Abdominal wall abscess (Infections and infestations) | 2 (2) | 0 (0)
Abscess intestinal (Infections and infestations) | 0 (0) | 1 (1)
Bronchopneumonia (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 1 (1)
Disseminated tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Empyema (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Peritoneal abscess (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 4 (4)
Postoperative wound infection (Infections and infestations) | 2 (2) | 2 (2)
Retroperitoneal abscess (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 3 (3) | 1 (1)
Septic shock (Infections and infestations) | 3 (3) | 0 (0)
Wound infection (Infections and infestations) | 10 (10) | 1 (1)
Rectal abscess (Infections and infestations) | 0 (0) | 1 (1)
Appendiceal abscess (Infections and infestations) | 0 (0) | 2 (2)
Haematoma infection (Infections and infestations) | 1 (1) | 1 (1)
Subdiaphragmatic abscess (Infections and infestations) | 0 (0) | 1 (1)
Abdominal infection (Infections and infestations) | 1 (1) | 1 (1)
Wound sepsis (Infections and infestations) | 0 (0) | 1 (1)
Wound abscess (Infections and infestations) | 0 (0) | 1 (1)
Abdominal abscess (Infections and infestations) | 2 (2) | 1 (1)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1)
Post procedural sepsis (Infections and infestations) | 1 (1) | 0 (0)
Failure to anastomose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Postoperative ileus (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound evisceration (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Postoperative respiratory distress (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural bile leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Anastomotic complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gastrointestinal disorder postoperative (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Intestinal anastomosis complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Chest X-ray abnormal (Investigations) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hairy cell leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Coma (Nervous system disorders) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Hemiplegia (Nervous system disorders) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 4 (4) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Shock (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Cardiovascular insufficiency (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Moxifloxacin (Avelox, BAY12-8039) (N=408) | Ertapenem (N=390)
Diarrhoea (Gastrointestinal disorders) | 23 (23) | 18 (18)
Nausea (Gastrointestinal disorders) | 30 (33) | 17 (18)
Wound infection (Infections and infestations) | 37 (37) | 28 (28)
Lipase increased (Investigations) | 25 (25) | 24 (24)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The agreed point of publication is 12/18 months after database lock at the earliest. Bayer will have up to 30/45 days to review publications and may request an additional publication delay of up to 60 days to allow for filing a patent application (if applicable). No publication of single center data should be done prior of publication if multi-center data.